CLINICAL TRIAL: NCT00698685
Title: Phase II Related or Unrelated Allogeneic Hematopoietic Cell Transplantation for High-Risk Malignancies, Using a Preparative Regimen of Pentostatin (Nipent®) and Alemtuzumab (Campath®)
Brief Title: Pentostatin and Alemtuzumab as a Preparative Regimen for Allogeneic Peripheral Blood Stem Cell Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Pentostatin/alemtuzumab regimen had greater risk of graft failure.
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-0624-04; R21CA106177 (NIH); 05110 (Other: University of Arizona); UARIZ-05-0624-01 (Other: University of Arizona); UARIZ-SRC17920 (Other: Arizona Cancer Center); NCT00543283 (obsolete NCT alias)
Record Dates: First submitted 2008-06-14; First posted 2008-06-17 (Estimated); Results first posted 2011-01-12 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Leukemia; Lymphoma; Hodgkin's Disease; Hematologic Neoplasms; Multiple Myeloma; Carcinoma, Renal Cell
Keywords: Allogeneic Hematopoietic Cell Transplantation; Preparative Regimen; Pentostatin; Alemtuzumab; Hodgkin Disease and Lymphoma, non-Hodgkin; leukemia, myeloid, acute; leukemia, lymphocytic, acute; leukemia, myeloid, chronic; leukemia, lymphocytic, chronic; Multiple Myeloma; Myelodysplastic Syndromes; Carcinoma, Renal Cell
MeSH Terms: conditions — Leukemia; Lymphoma; Hodgkin Disease; Hematologic Neoplasms; Multiple Myeloma; Carcinoma, Renal Cell; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Lymphocytic, Chronic, B-Cell; Myelodysplastic Syndromes | interventions — Pentostatin; Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Preparative Regimen (Experimental): Days - 8 through -6: pentostatin 4 mg/m2/24 hr as a continuous intravenous infusion (CIVI) (total cumulative dose, 12 mg/m2 over 3 days)
  Days - 5 through - 1: alemtuzumab 20 mg per dose intravenously over 8 hours daily for 5 doses (total cumulative dose, 100 mg)
  Followed by Allogeneic hematopoietic stem cell transplantation, related or unrelated donor, on day 0. Patients also receive cyclosporine intravenous (IV) continuously beginning on day -2, continuing (IV or orally) until day 100, followed by a taper.
  Interventions: Drug: Pentostatin; Biological: Alemtuzumab; Procedure: Allogeneic hematopoietic stem cell transplantation

INTERVENTIONS:
Drug: Pentostatin — Days - 8 through -6: pentostatin 4 mg/m2/24 hr as a continuous intravenous infusion (CIVI) (total cumulative dose, 12 mg/m2 over 3 days)
  Other Names: Nipent
Biological: Alemtuzumab — Days - 5 through - 1: alemtuzumab 20 mg per dose intravenously over 8 hours daily for 5 doses (total cumulative dose, 100 mg)
  Other Names: Campath
Procedure: Allogeneic hematopoietic stem cell transplantation — Infusion of related or unrelated donor peripheral blood progenitor cells on day 0.
  Other Names: HSCT

SUMMARY:
This study tests the hypothesis that a purely immunosuppressive preparative regimen allows engraftment of related or unrelated allogeneic hematopoietic stem cells in subjects with high-risk malignancies, without causing the post-transplant myelosuppression (e.g., neutropenia, thrombocytopenia) that occurs with currently used reduced-intensity (nonmyeloablative) preparative regimens. This study incorporates both safety and efficacy endpoints and evaluates a novel preparative regimen of alemtuzumab plus continuous-infusion pentostatin, two immunosuppressive agents with different mechanisms of action, in recipients of related or unrelated allogeneic hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
Primary Objectives of the study:

* To determine the efficacy of a preparative regimen of pentostatin and alemtuzumab plus related or unrelated allogeneic peripheral blood stem cell transplantation (PBSCT) in inducing durable donor lymphohematopoietic cell chimerism (defined as at least 50% donor cells in the peripheral blood) by 100 days after PBSCT (day +100) in subjects with high-risk malignancies who are at high risk for morbidity and mortality with conventional intensive pre-transplant conditioning regimens.
* To determine the safety of a preparative regimen of pentostatin and alemtuzumab plus related or unrelated allogeneic PBSCT, as measured by the non-relapse mortality at day +100 in the study subject population.

ELIGIBILITY:
Inclusion Criteria:

One of these diagnoses:

* Acute myeloid leukemia in complete or partial remission
* Acute lymphocytic leukemia in complete or partial remission
* Chronic myeloid leukemia in first or subsequent chronic phase or accelerated phase
* Chronic lymphocytic leukemia that has recurred or failed after at least one course of front-line therapy
* Hodgkin's disease or non-Hodgkin's lymphoma that has failed front-line therapy, is in second or subsequent remission, or is in chemosensitive relapse
* Multiple myeloma that is in complete or partial remission or in chemosensitive relapse
* Myelodysplastic Syndrome classified as intermediate-2 or high risk according to International Prognostic Scoring System
* Metastatic renal cell carcinoma that has failed at least one previous front-line chemotherapy and/or biological therapy regimen and that is radiographically detectable and evaluable
* Treatment with at least one previous course of chemotherapy or biological therapy for the malignancy for which allogeneic PBPCT is being considered (i.e., a subject cannot be enrolled on this study for initial treatment of a malignancy).

AND at least one of the following:

* Age 50 years or older.
* Previous transplant with autologous or allogeneic hematopoietic cells (peripheral blood, bone marrow, or placental blood).
* High-risk status of hematologic malignancy, i.e., not in first complete remission or first chronic phase.
* Presence of other medical condition that could place subject at unacceptably high risk of regimen-related mortality such as documented chronic bronchitis or emphysema; decreased cardiac ejection fraction (but with ejection fraction at least 30%), or history of coronary artery disease; renal insufficiency (but with creatinine clearance at least 30 mL/min); hepatic cirrhosis (but with normal hepatic synthetic function); or documented or presumed invasive fungal infection requiring treatment with intravenous antifungal agent(s).

Exclusion Criteria:

* Eligibility for another clinical therapeutic protocol or standard-of-care treatment that offers higher probability of cure or long-term control of subject's malignancy.
* Progressive Hodgkin's disease, non-Hodgkin's lymphoma, Hodgkin disease or multiple myeloma that is refractory to salvage chemotherapy.
* Acute leukemia (AML or ALL) in relapse, CML in blast phase/blast crisis, or MDS with greater than 30% marrow involvement (MDS-AML). Subjects with these disease characteristics may be considered for this study if complete or partial remissions (CRs or PRs) occur after salvage chemotherapy.
* Severe organ dysfunction, such as: cardiac ejection fraction below 30% or symptomatic ischemic cardiac disease; creatinine clearance below 30 mL/min; carbon monoxide diffusing capacity (DLCO) below 35% and/or need for supplemental oxygen; severe hepatic cirrhosis with ascites and/or varices; hepatic dysfunction associated with abnormal synthetic function (e.g., coagulopathy) and/or bilirubin greater than two times upper limit of normal and/or transaminases (AST or ALT) above four times upper limit of normal.
* Untreated or progressive central nervous system involvement by malignancy
* Subject is pregnant or breast-feeding.
* Karnofsky score below 50
* Seropositivity for human immunodeficiency virus (HIV).
* Life expectancy less than 12 weeks with conventional treatments.
* For subjects who are fertile, refusal to practice contraception upon entering this study and for at least 12 months after PBPCT or after cessation of immunosuppressive treatments (e.g., cyclosporine), whichever occurs later.
* Failure to obtain at least 5.0 x 106 allogeneic donor CD34+ cells per kg of recipient weight in PBPC product.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2006-01-23 (Actual); Primary Completion 2009-04-13 (Actual); Study Completion 2011-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Yeager, MD, Principal Investigator — University of Arizona
Locations (2):
- United States (2):
  - Arizona Cancer Center at UMC North/University Medical Center, Tucson, Arizona
  - Arizona Cancer Center at UMC North, Tucson, Arizona

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Following University of Arizona IRB review and approval, the study opened to accrual on November 2005 at the Arizona Cancer Center clinic and University Medical Center sites [Tucson, Arizona].
Pre-assignment Details: Following consent process, subjects who consented to participate were screened per the selection criteria in the study.
Groups:
- Preparative Regimen of Pentostatin and Alemtuzumab: Pentostatin and Alemtuzumab as a Preparative Regimen for Allogeneic [related or unrelated] Hematopoietic SCT.
  Pentostatin: 4 mg/m2/24 hour IV continuously over 72 hours on days -8 to -6. Alemtuzumab: 20 mg per dose IV over 8 hours on days -5 to -1. Patients then received infusion of related or unrelated donor peripheral blood progenitor cells on day 0. Patients also receive cyclosporine IV continuously beginning on day -2, continuing (IV or orally) until day 100, followed by a taper.
Period: Overall Study
Arm/Group | Preparative Regimen of Pentostatin and Alemtuzumab
Started | 14
Completed | 12
Not Completed | 2
Not completed — Sister withdrew as donor | 1
Not completed — Off study pre transplant by clinic MD | 1

BASELINE CHARACTERISTICS:
Arm/Group | Preparative Regimen of Pentostatin and Alemtuzumab
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Actuarial Probability of Donor Hematopoietic Engraftment (Defined as at Least 50% Donor DNA in Bone Marrow at Day 100).
Description: The number of participants with donor hematopoietic engraftment at day 100 is reported in the data table, and the actuarial probability is calculated using the Kaplan-Meier product-limit estimate statistic, as reported in the statistical analysis section below.
Time Frame: Day 100 after transplant.
Population: All participants who completed treatment and underwent allogeneic transplant.
Measure: Number; unit: participants
Arm/Group | Preparative Regimen of Pentostatin and Alemtuzumab
Number analyzed (Participants) | 12
participants | 4
Statistical Analysis 1: Comparison: Preparative Regimen of Pentostatin and Alemtuzumab; Test type: Superiority or Other; actuarial probability of engraftment = 70 — Actuarial probability of engraftment at day +100 is calculated according to the product-limit estimate method

2. Primary Outcome: Non-relapse Mortality at or Before Day 100
Description: The primary safety outcome is indicated by the number of participants who died at or before Day 100 after transplant for any reason other than relapse of disease (Leukemia, Lymphoma, Hodgkin's disease, Hematologic Neoplasms, Multiple Myeloma, Renal Cell Carcinoma).
Time Frame: Day 100 after transplant
Population: All participants who received at least 1 day of treatment.
Measure: Number; unit: Participants
Arm/Group | Preparative Regimen of Pentostatin and Alemtuzumab
Number analyzed (Participants) | 13
Participants | 3

ADVERSE EVENTS:
Time Frame: Adverse event data for this study was collected from January 23, 2006 to April 13, 2009.
Description: Adverse event data was collected and entered into the AZCC database which is password protected. The safety population is defined to be all participants who completed at least 1 day of treatment.
Arm/Group | Preparative Regimen of Pentostatin and Alemtuzumab
Serious Adverse Events (participants affected / at risk) | 8/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preparative Regimen of Pentostatin and Alemtuzumab (N=13)
metabolic/laboratory: elevated AST and ALT (Blood and lymphatic system disorders) | 1 (1) — These blood chemistries returned to normal within several days after cessation of pentostatin infusion and without specific intervention: probably associated with the infusion of pentostatin.
hemorrhagic cystitis associated with BK virus (Renal and urinary disorders) | 1 (1) — Developed about 50 days after unrelated PBPCT;required hospital stay for continuous bladder irrigation and transfusions of red cells and platelets; also had elective cystoscopy, at which time clot was evacuated from the bladder. Possibly related.
hypoxia and dyspnea which was a result of pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Occurred without evidence of donor engraftment. subject had comorbidities [i.e., coronary artery disease] died with multisystem failure. Assessed as expected SAE and was possibly related.
altered mental status and progressive obtundation [disseminated toxoplasmosis] (Infections and infestations) | 1 (1) — After extensive evaluation, determined subject had disseminated toxoplasmosis. Subject died shortly after initiation of definitive therapy for toxoplasmosis. Assessed expected SAE [infections] and possibly related to investigational treatment.
hyperbilirubinemia (Blood and lymphatic system disorders) | 1 (1) — Due to progressive hepatic infiltration by Hodgkin's disease and felt to be an expected SAE that was related to subject's aggressive underlying malignancy and unrelated to investigational treatment.
disseminated toxoplasmosis (Infections and infestations) | 1 (1) — Subject had persistent fevers and disseminated toxoplasmosis determined by quantitative PCR on a blood sample. Assessed as expected SAE (infections)and possibly related to investigational treatment.
thrombotic microangiopathy (Renal and urinary disorders) | 1 (1) — Developed in May 2009 about 6 months after administration of investigational treatment and required hemodialysis. Assessed as expected SAE and unrelated to the investigational treatment.
Death on study, post BMT (Cardiac disorders) | 1 (1) — Cardiac and respiratory failure.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preparative Regimen of Pentostatin and Alemtuzumab (N=13)
Blood/Bone Marrow (Blood and lymphatic system disorders) | 5 (63)
DIC (disseminated intravascular coagulation) (Blood and lymphatic system disorders) | 1 (1)
Cardiac General (Cardiac disorders) | 6 (10)
Cardiac Arrhythmia (Cardiac disorders) | 1 (1)
Edema: limb (Blood and lymphatic system disorders) | 4 (9)
Edema: viscera (Blood and lymphatic system disorders) | 1 (1)
Fibrinogen (Blood and lymphatic system disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 8 (36)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 4 (8)
Lymphatics (Blood and lymphatic system disorders) | 8 (17)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 7 (35)
PTT (Partial Thromboplastin Time) (Blood and lymphatic system disorders) | 2 (2)
Cardiac troponin T (cTnT) (Cardiac disorders) | 1 (2)
Hypertension (Cardiac disorders) | 5 (7)
Hypotension (Cardiac disorders) | 4 (5)
Pericardial effusion (non-malignant) (Cardiac disorders) | 1 (1)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 2 (4)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)
Death not associated with CTCAE term (Eye disorders) | 1 (1)
Ocular/Visual (Eye disorders) | 3 (4)
Vision-photophobia (Eye disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 3 (7)
Constipation (Gastrointestinal disorders) | 4 (9)
Dehydration (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (3)
Flatulence (Gastrointestinal disorders) | 1 (2)
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 1 (1)
Gastrointestinal (Gastrointestinal disorders) | 6 (33)
Heartburn/dyspepsia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (22)
Vomiting (Gastrointestinal disorders) | 5 (12)
Constitutional Symptoms (General disorders) | 7 (33)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 4 (5)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC >1.0 x="" 10e9=""/L) (General disorders) | 6 (13)
Insomnia (General disorders) | 4 (10)
Pain (General disorders) | 12 (98)
Rigors/chills (General disorders) | 5 (7)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 2 (2)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 2 (2)
Allergy/Immunology (Immune system disorders) | 3 (6)
Autoimmune reaction (Immune system disorders) | 1 (2)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 2 (2)
Infection (Infections and infestations) | 8 (20)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 1 (1)
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 1 (2)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 3 (12)
Alkaline phosphatase, increased (Metabolism and nutrition disorders) | 1 (1)
ALT, SGPT (serum glutamic pyruvic transaminase), increased (Metabolism and nutrition disorders) | 6 (8)
AST, SGOT(serum glutamic oxaloacetic transaminase), increased (Metabolism and nutrition disorders) | 6 (7)
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 2 (10)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 2 (2)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 2 (4)
Creatinine, increased (Metabolism and nutrition disorders) | 6 (18)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 4 (36)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 7 (40)
Metabolic/Laboratory (Metabolism and nutrition disorders) | 10 (84)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 2 (3)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 1 (1)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 7 (19)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 3 (5)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 1 (1)
Musculoskeletal/Soft Tissue (Musculoskeletal and connective tissue disorders) | 2 (2)
Confusion (Nervous system disorders) | 2 (3)
Dizziness (Nervous system disorders) | 1 (1)
Extrapyramidal/involuntary movement/restlessness (Nervous system disorders) | 1 (1)
Mood alteration (Nervous system disorders) | 4 (10)
Neurology (Nervous system disorders) | 6 (14)
Neuropathy: sensory (Nervous system disorders) | 1 (1)
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Bladder spasms (Renal and urinary disorders) | 1 (1)
Cystitis (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 4 (7)
Renal/Genitourinary (Renal and urinary disorders) | 5 (7) — Hematuria, anuria, renal insufficiency, urinary tract infection.
Urinary frequency/urgency (Renal and urinary disorders) | 1 (1)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (7)
Hemorrhage, pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hemorrhage/Bleeding (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pulmonary/Upper Respiratory (Respiratory, thoracic and mediastinal disorders) | 7 (28)
Cytokine release syndrome/acute infusion reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatology/Skin (Skin and subcutaneous tissue disorders) | 8 (18)
Flushing (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 2 (2)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1)
Rash: erythema multiforme (e.g., Stevens-Johnson syndrome, toxic epidermal necrolysis) (Skin and subcutaneous tissue disorders) | 1 (1)
Hemorrhage/Bleeding (Surgical and medical procedures) | 2 (3)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 1 (2)
Vascular (Vascular disorders) | 4 (5) — Increased [cyclosporine] CSA level, jugular venous distention, port occlusion [2].

LIMITATIONS AND CAVEATS:
We did not meet criteria to stop the study because of nonrelapse mortality (safety endpoint). However, we stopped accrual to the study because of failure to meet minimal criteria for engraftment (efficacy endpoint).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes